CLINICAL TRIAL: NCT04174950
Title: Effect of Perioperative ERAS Based Nursing Intervention on Hope Level of Patients With Laryngeal Cancer
Brief Title: Perioperative ERAS Based Nursing Intervention for Laryngeal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, yuxuefei, Head Nurse, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-107
Record Dates: First submitted 2019-07-12; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Laryngeal Cancer; Nursing
Keywords: Laryngeal cancer; enhanced recovery after surgery; hope level
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants were allocated into two groups randomly.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Routine perioperative nursing intervention
  Interventions: Other: Routine nursing care
- experimental group (Experimental): Perioperative ERAS Based Nursing Model
  Interventions: Other: Perioperative Enhanced Recovery After Surgery (ERAS) Based Nursing Model

INTERVENTIONS:
Other: Routine nursing care — routine perioperative nursing intervention, including intensive observation of vital signs, preoperative education, postoperative communication and instruction on diet. NPO after the dinner one day before operation. Patients are instructed to NPO 3 days after surgery and patients should stay on the bed for 3 days. Urinary catheter is always kept for 48 hours or more.
  Arms: control group
Other: Perioperative Enhanced Recovery After Surgery (ERAS) Based Nursing Model — Establish ERAS nursing team and formulate ERAS nursing intervention. Nothing by mouth (NPO) 6 hours before operation and no water 4 hours before operation. Patients are given fluid food 24 hours after surgery. Urinary catheter is removed within 24 hours after surgery and encourage patient to mobile 24 hours after surgery. Give support to pain control and psychological support. Intensive observation of vital signs, preoperative education, postoperative communication and instruction on diet were also given to patients.
  Arms: experimental group

SUMMARY:
To explore the effect of perioperative ERAS based nursing model on the hope level and recovery of patients with laryngeal cancer.

DETAILED DESCRIPTION:
200 patients who were diagnosed with laryngeal cancer and received total or partial laryngectomy were included. They were allocated into experimental and control group. Patients in experimental group were given ERAS based nursing intervention. Control group were given routine nursing intervention. Compare hope level, postoperative recovery, complication between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients were confirmed as laryngeal cancer by CT scan.
* Patients were given total or partial laryngectomy.

Exclusion Criteria:

* Unconscious or psychiatric patients.
* Patients with distant metastasis or recurrence of cancer
* Patients with coagulation dysfunction
* Patients with severe cardiac, hepatic or renal dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Hope level | the day before surgery
  Herth Hope Index which have 12 items. Each item is rated from 1 to 4. Score 1 represents lowest level. Score 4 represents highest level. Total score is 48.
Hope level | Day 10 after surgery
  Herth Hope Index which have 12 items. Each item is rated from 1 to 4. Score 1 represents lowest level. Score 4 represents highest level. Total score is 48.

SECONDARY OUTCOMES:
Ambulation time | Day 3 after surgery
  record the time of first ambulation
Level of Pain | Day 3 after surgery
  Numerical rating scale is a common pain rating scale. The score ranges from 0 to 10. 0 is no pain, 10 is the most severe pain.
Postoperative complication | Day 30 after surgery
  incidence of infection, malnutrition and Viscosity of sputum
Length of stay | Day 30 after surgery
  the days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Yu, bachelor, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No